CLINICAL TRIAL: NCT07136181
Title: A Multicenter Phase Ib/II Study to Evaluate the Safety, Efficacy and Pharmacokinetics of NBM-BMX in Patients With Metastatic Uveal Melanoma
Brief Title: Evaluation of the Safety, Efficacy, and Pharmacokinetics of NBM-BMX in Patients With Metastatic Uveal Melanoma
Acronym: NBM-BMX-UM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novelwise Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBM-BMX-004; IND177628 (Registry Identifier: FDA)
Record Dates: First submitted 2025-07-15; First posted 2025-08-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Uveal Melanoma; Uveal Melanoma, Metastatic; Uveal Melanoma, Recurrent; Eye Cancer, Intraocular Melanoma; Eye Cancer
Keywords: Metastatic Uveal Melanoma; Uveal Melanoma; Eye Cancer; Intraocular Melanoma; Choroidal Melanoma; NBM-BMX; Histone Deacetylase Inhibitor (HDAC inhibitor); Phase 1b/2 Study; Pharmacokinetics
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis; Recurrence; Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- In the present Phase Ib/II study, up to three dose levels are planned (Experimental): NBM-BMX is a small molecule inhibitor of HDAC8 currently in Phase I testing that has demonstrated activity in a metastatic UM patient. Given the role of the HDAC8 pathway on development and growth of uveal melanoma and the initial clinical activity in the UM setting, there is a high probability that NBM-BMX would have efficacy in this disease
  In the present Phase Ib/II study, up to four dose levels are planned:
  * Dose Level 1: 200 mg daily (100 mg BID)
  * Dose Level 2: 400 mg daily (200 mg BID)
  * Dose Level 3: 600 mg daily (300 mg BID)
  * Dose Level 4: 800 mg daily (400 mg BID) A total daily dose of 600 mg (300 mg BID) of the NBM-BMX dry powder formulation has been well tolerated in patients with advanced solid tumors. As three subjects have completed treatment at this dose level without evidence of DLTs, the 200 mg/day dose selected for this trial represents two full dose levels below the highest tolerated dose and is expected to be both safe and pharmacologically active.
  Interventions: Drug: NBM-BMX Capsule are proprietary products developed by Novelwise Pharmaceutical Corporation (Novelwise) for treatment of patients suffering from cancers.

INTERVENTIONS:
Drug: NBM-BMX Capsule are proprietary products developed by Novelwise Pharmaceutical Corporation (Novelwise) for treatment of patients suffering from cancers. — NBM-BMX is a small molecule inhibitor of HDAC8. The majority of metastasizing uveal melanoma (UM) cases are characterized by the presence of BAP1 mutations. However, as BAP1 mutations lead to a loss of function, therapeutic strategies have primarily focused on exploiting vulnerabilities resulting from BAP1 loss or targeting downstream effectors affected by the BAP1-deficient phenotype. In uveal melanocytes, the absence of BAP1 disrupts their differentiated cell identity, potentially contributing to the metastatic behavior observed in BAP1-mutant UM cells. This differentiation block in the melanocytic lineage is thought to be influenced, at least in part, by the activation of HDAC8 downstream, which leads to the repression of differentiation genes through acetylation of the histone H3K27 at the promoter and enhancers associated with these genes. Consequently, inhibiting HDAC8 could potentially reverse the differentiation block caused by the loss of BAP1.

SUMMARY:
This study is being done to find the best dose of an investigational drug called NBM-BMX for people with metastatic uveal melanoma, a type of eye cancer that has spread to other parts of the body.

The study will help doctors learn about the side effects of NBM-BMX, how the drug is processed in the body, and whether it may slow down or shrink tumors.

Participants will take NBM-BMX as a capsule by mouth twice daily on an empty stomach with at least six ounces (180 mL) of water. No food or drink (other than water) should be consumed for at least two hours after each dose.

Participants will visit the clinic about once every week or two for exams and blood tests while taking NBM-BMX. After stopping treatment, a follow-up visit will occur about 30 days later.

Treatment may continue as long as the cancer does not get worse and side effects remain manageable.

DETAILED DESCRIPTION:
NBM-BMX will be administered orally twice daily (BID) at approximately 12 ± 2-hour intervals for 28 consecutive days per cycle, beginning on Day 1 of Cycle 1. Patients will continue treatment until disease progression, intolerable toxicity likely attributable to NBM-BMX, or voluntary withdrawal from the study. If disease progression is equivocal and, in the investigator's judgment, the patient appears to be benefiting, treatment may continue with close monitoring and re-evaluation at the next scheduled tumor assessment.

The study drug will be provided in 100 mg dry powder hard gel capsules. All dosing will be performed on an outpatient basis. NBM-BMX must be taken on an empty stomach with at least six ounces (180 mL) of water.

Patients should not eat food for at least 1 hour before and 2 hours after each dose of NBM-BMX. Only water is permitted during this fasting window.

To minimize the risk of altered absorption, other oral medications should be taken at least 1 hour before or 2 hours after NBM-BMX administration, unless otherwise approved by the Investigator.

Due to the pH-dependent solubility of NBM-BMX, acid-reducing agents (such as PPIs or H2 blockers) may reduce drug absorption. Patients must avoid taking these agents during the study. Local antacids may be taken at least 2 hours before or after dosing if clinically indicated.

Compliance with these fasting instructions should be reinforced at each clinic visit and documented in the patient diary and/or source records.

At each study visit, patients will be dispensed enough drug for daily dosing until the next visit, along with specific instructions on the number of capsules to take in the morning and evening. Drug accountability, including the number of capsules and containers dispensed, patient number, and date of dispensing, will be recorded in the Case Report Form. Patients must store the drug in the original container at room temperature (15 to 25°C) in a secure location away from excessive heat or moisture. Participants will be instructed not to remove or consume the desiccant included in each bottle.

Prior to dispensing, all women of childbearing potential must have a negative pregnancy test, be counseled on the teratogenic potential of NBM-BMX, and agree to use two acceptable forms of contraception, including one barrier method. If pregnancy is suspected, dosing must be discontinued immediately. If pregnancy is confirmed by serum test, the patient will be withdrawn from the study and complete the early termination visit. If pregnancy is ruled out, treatment may be resumed.

Patients will be instructed to complete a dosing diary, recording the date and time of each dose, any missed doses, and any symptoms or side effects experienced. Research staff will review the diary, address any concerns, and collect unused medication and empty containers at each study visit. Every effort will be made to retrieve all dispensed containers; if unsuccessful, the reason will be documented. If a patient misses a dose, participants should not attempt to make it up and should resume treatment at the next scheduled time. All missed doses must be documented in the dosing diary.

SCREENING AND PRETREATMENT ASSESSMENTS Screening tests and evaluations will be used to determine the eligibility of each patient for study inclusion. All patients must provide written informed consent before any study-specific procedures and assessments are performed and any exclusionary medications are discontinued for the purposes of establishing eligibility. Screening evaluations will be performed within the 14 days preceding Day 1, unless otherwise specified. Results of tests or examinations performed as standard of care prior to obtaining informed consent and within 14 days prior to study entry may be used rather than repeating required tests.

ASSESSMENTS DURING TREATMENT All visits must occur within ± 3 days from the scheduled date, unless otherwise noted. All assessments will be performed on the day of the specified visit unless a time window is specified. Assessments scheduled on the day of study drug administration (Day 1) of each cycle should be performed prior to study drug administration, unless otherwise noted.

STUDY COMPLETION/EARLY TERMINATION VISIT Patients who discontinue from the study will be asked to return to the clinic within 30 days of the last dose of NBM-BMX for a follow-up visit.

Assessments and Endpoints Safety will be assessed through adverse event monitoring, vital signs, physical examinations, ECGs, and clinical laboratory tests. Pharmacokinetics will be evaluated at predefined time points. Tumor response will be assessed using RECIST 1.1 criteria every 8 weeks during treatment.

Expanded Access Information:

An Expanded Access program for this investigational product (NBM-BMX) is available for eligible patients under FDA regulations.

For more information, please contact expandedaccess@novelwisepharma.com or visit our website at www.novelwiseoncology.com/expanded-access

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet the following criteria to be eligible for study entry:

1. Signed, written IRB-approved informed consent.
2. Men and women age ≥ 18 years
3. ECOG Performance status ≤ 2
4. Have measurable disease based on RECIST 1.1
5. Histologic or cytologic confirmation of metastatic uveal melanoma
6. Previous Therapy

   * Surgery: Previous surgery is permitted provided that a minimum of 28 days (4 weeks) has elapsed between any major surgery and date of registration, and that wound healing has occurred.
   * Cytotoxic Chemotherapy: There is no limit to the number of prior regimens received.
   * Other Systemic Therapy: There is no limit to the number of prior therapies received for metastatic uveal melanoma. Prior treatment with tebentafusp is required for HLA-A*02:01-positive patients unless unavailable or clinically inappropriate, as determined by the investigator. Prior HDAC inhibitor treatment is not permitted.

   Patients must have recovered (to baseline or ≤ grade 1) from all reversible toxicity related to prior chemotherapy or systemic therapy and have adequate washout as follows:

   Longest of one of the following:
   * Two weeks,
   * 5 half-lives for investigational agents,

     o For anti-cancer therapies with half-lives > 8 days, a washout period of at least 28 days will be acceptable,
   * Standard cycle length of standard therapies.
7. QTcF <= 480 msec
8. Adequate hematopoietic capacity, as defined by the following:

   * Hemoglobin ≥ 9.0 g/dL and not transfusion dependent
   * Platelets ≥ 100,000/mm3
   * Absolute neutrophil count ≥ 1,500 cells/mm3
9. Adequate hepatic function, as defined by the following:

   * AST and ALT ≤ 2.5 times upper limit of normal (ULN) or ≤ 5 times ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 x ULN or within 3x the ULN for patients with Gilbert disease
   * Albumin ≥ 3.0 g/dL
10. Adequate renal function, as defined by the following:

    - Renal: calculated creatinine clearance >45 mL/min for patients between 18 and 70 years old with abnormal, increased, creatinine levels (Cockcroft-Gault formula; Appendix F). For patients who are greater than 70 years old, investigator judgment may be used to assess the renal risk of study participation.
11. Women/men of childbearing potential must have agreed to use two effective contraceptive methods while on study and for 6 months after the last dose of NBM-BMX.
12. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

Patients who meet the following criteria will be excluded from study entry:

1. Pregnant or nursing women. NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation and for at least 6 months after the last dose of NBM-BMX. Should a man father a child, or a woman become pregnant or suspect she is pregnant while participating in this study, he or she should inform the treating physician immediately.
2. Concurrent non-protocol-specified anti-tumor therapy (e.g., chemotherapy, other targeted therapy, radiation therapy, or photodynamic therapy)
3. History of other malignancies within 3 years of Day 1, except for tumors with a negligible risk for metastasis or death, such as adequately treated squamous-cell carcinoma of the skin, ductal carcinoma in situ of the breast, or carcinoma in situ of the cervix.
4. Active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
5. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk from treatment complications.
6. Difficulty with swallowing oral medications.
7. Currently taking moderate and strong inhibitors (e.g., gemfibrozil) or inducers of CYP2C8.
8. A positive test for hepatitis B (HBsAg) and/or hepatitis C (anti-HCV antibody), unless the HBV DNA level and/or HCV RNA level is below the limit of detection.
9. Any of the following within 3 months of the first dose of NBM-BMX: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack.
10. Current use or anticipated need for P-gp or BCRP inhibitors during the study period.
11. Use of proton pump inhibitors (PPIs), H2-receptor antagonists, or other systemic acid-reducing agents within 7 days prior to Cycle 1 Day 1 or planned use during the study treatment period, unless the patient can be switched to local antacids (e.g., calcium carbonate or aluminum hydroxide) taken at least 2 hours before or after NBM-BMX dosing.

Patients unable or unwilling to comply with this restriction should be excluded. Exceptions must be discussed with and approved by the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-03-28 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of dose-limiting toxicities (DLTs) | Time Frame: Cycle 1 (up to 28 days)
  Participants experiencing a DLT during Cycle 1 (28 days)
Phase Ib: Maximum Tolerated Dose (MTD) | Cycle 1 (up to 28 days)
  The highest dose level with ≤1 of 6 participants with a DLT, based on the incidence of DLTs at each dose level of NBM-BMX during Cycle 1 (28 days). MTD will inform the recommended Phase 2 dose (RP2D) of NBM-BMX
Phase II: Objective Response Rate (ORR) | Assessed every 8-12 weeks from first dose; up to ~24 months
  Proportion of patients with complete response (CR) + partial response (PR) determined per RECIST 1.1 while on NBM-BMX.

SECONDARY OUTCOMES:
Phase Ib: Safety and Tolerability | From first dose through 30 days after last dose (up to ~25 months)
  Incidence, severity, and type of adverse events graded per NCI CTCAE v5.0
Phase Ib: Objective Response Rate (ORR) | Assessed every 8 -12 weeks from first dose; up to ~24 months
  Percentage of participants with confirmed Complete Response (CR) or Partial Response (PR) per RECIST v1.1.
Phase Ib. PK: Maximum plasma concentration (Cmax) | Cycle 1 Day 1: pre-dose to 12 hours post-dose
  Cmax of NBM-BMX from plasma concentration-time profile (suggested unit: ng/mL)
Phase Ib. PK: Time to Cmax (Tmax) | Cycle 1 Day 1: pre-dose to 12 hours post-dose
  Tmax of NBM-BMX from plasma concentration-time profile (unit: hours)
Phase Ib. PK: Area under the curve (AUC 0-12) | Cycle 1 Day 1: pre-dose to 12 hours post-dose
  AUC from 0 to 12 hours after the morning dose (unit: ng·h/mL)
Phase Ib. PK: Elimination half-life (T½) | Cycle 1 Day 1
  Terminal plasma half-life derived from concentration-time profile (unit: hours)
Phase Ib. PK: Apparent oral clearance (CL/F) | Cycle 1 Day 1
  CL/F from non-compartmental analysis (unit: L/h)
Phase Ib. PK: Apparent volume of distribution (Vd/F) | Cycle 1 Day 1
  Vd/F from non-compartmental analysis (unit: L)
Phase II: 3-Month Progression-Free Survival (PFS) Rate | 3 months from treatment initiation
  Proportion of participants alive and progression-free at 3 months per RECIST v1.1.
Phase II: Overall Survival (OS) | Up to ~24 months
  Time from first dose to death from any cause

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Honor Health Resarch Institute, Scottsdale, Arizona
  - Sarah Cannon Research Institute (SCRI) - Denver HealthONE Location, Denver, Colorado
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Char DH, Kroll SM, Castro J. Ten-year follow-up of helium ion therapy for uveal melanoma. Am J Ophthalmol. 1998 Jan;125(1):81-9. doi: 10.1016/s0002-9394(99)80238-4. PMID 9437317
- [Result] Yang W, Feng Y, Zhou J, Cheung OK, Cao J, Wang J, Tang W, Tu Y, Xu L, Wu F, Tan Z, Sun H, Tian Y, Wong J, Lai PB, Chan SL, Chan AW, Tan PB, Chen Z, Sung JJ, Yip KY, To KF, Cheng AS. A selective HDAC8 inhibitor potentiates antitumor immunity and efficacy of immune checkpoint blockade in hepatocellular carcinoma. Sci Transl Med. 2021 Apr 7;13(588):eaaz6804. doi: 10.1126/scitranslmed.aaz6804. PMID 33827976
- [Result] Diener-West M, Reynolds SM, Agugliaro DJ, Caldwell R, Cumming K, Earle JD, Hawkins BS, Hayman JA, Jaiyesimi I, Jampol LM, Kirkwood JM, Koh WJ, Robertson DM, Shaw JM, Straatsma BR, Thoma J; Collaborative Ocular Melanoma Study Group. Development of metastatic disease after enrollment in the COMS trials for treatment of choroidal melanoma: Collaborative Ocular Melanoma Study Group Report No. 26. Arch Ophthalmol. 2005 Dec;123(12):1639-43. doi: 10.1001/archopht.123.12.1639. PMID 16344433